CLINICAL TRIAL: NCT05856591
Title: Delivering Food Resources & Kitchen Skills (FoRKS) to Adults With Food Insecurity and Hypertension: An RCT
Brief Title: Delivering Food Resources & Kitchen Skills (FoRKS) to Adults With Food Insecurity and Hypertension
Acronym: FoRKS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Daniel Clark, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16773; R01MD017961 (NIH)
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Food Insecurity; Hypertension; Nutrition; Disease Management
Keywords: randomized controlled trial; kitchen skills; diet; social determinants of health
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (EUC) (Active Comparator): Participants randomized to EUC will have access to existing usual primary care services. They will also be enrolled in Hypertension Self-Management Education and Support (SMES) class ("Hypertension group"), which is an existing CDC-endorsed program offered at Eskenazi Health to provide information and skills for managing hypertension (HTN). Classes are led by registered dietitians via Webex.
  Interventions: Behavioral: Enhanced Usual Care (EUC)
- Food Resources & Kitchen Skills (FoRKS) (Experimental): Participants randomized to FoRKS will attend weekly HTN SMES classes separately from EUC participants. SMES classes will include the EUC curriculum stated above and an introduction to the upcoming FoRKS intervention.
  Following HTN SMES completion, FoRKS continues with home-delivered Mediterranean-style ingredient kits, food management lessons, and hands-on cooking classes in one's own kitchen. Classes are led by registered dietitians via Webex. Classes are held twice per week thru Week 12, then only once per week through Week 16.
  Interventions: Behavioral: Food Resources & Kitchen Skills (FoRKS)

INTERVENTIONS:
Behavioral: Food Resources & Kitchen Skills (FoRKS) — Food Resources & Kitchen Skills (FoRKS) includes 5 weeks of hypertension classes followed by 11 weeks of home-delivered Mediterranean-style ingredient kits and virtual cooking classes with embedded lessons in kitchen organization, tool use, nutrition, budgeting, and shopping.
  Arms: Food Resources & Kitchen Skills (FoRKS)
Behavioral: Enhanced Usual Care (EUC) — Enhanced Usual Care (EUC) includes 5 weeks of hypertension classes.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The goal of this clinical trial is to determine the impact of a home-delivered foods and kitchen skills program on health and nutrition in adults with high blood pressure and food insecurity.

Researchers will compare Food Resources & Kitchen Skills (FoRKS) and Enhanced Usual Care (EUC) to evaluate the effects on mean systolic blood pressure (SPB), HbA1c, food security and nutrition.

Participants will complete 24-hr blood pressure monitoring, standard blood pressure measurements, weight, finger stick for A1c point-of-care testing, and questionnaires.

DETAILED DESCRIPTION:
This behavioral randomized controlled trial will evaluate nutritious food delivery and cooking classes (FoRKS) versus enhanced usual care (EUC) in adults with food insecurity and systolic blood pressure of ≥120 mm Hg. This project seeks to evaluate the potential for hands-on training in food management skills to create lasting improvements in food security, self-efficacy, nutrition, and risk factor reduction in persons with prevalent chronic disease.

Adults who pass the telephone screen will be invited to complete a blood pressure check for final eligibility determination. Participants must receive an average systolic read of ≥120 mmHG across 3 standard BP readings with designated wait periods; a maximum of 5 readings may be attempted to receive 3 successful measurements necessary to calculate the average. Participants who meet criteria and give informed consent will complete a full baseline assessment consisting of questionnaires, finger stick for A1c point-of-care testing, weight, and 24-hour ambulatory blood pressure before randomization to one of two arms:

1. Enhanced Usual Care (EUC), consisting of access to existing usual primary care services such as social determinants of health screenings, referrals to food pantries, and assistance enrolling in food assistance programs. They will be enrolled in a 5-week Hypertension Self-Management Education and Support (SMES) class, which is an existing CDC-endorsed program offered at Eskenazi to provide information and skills for managing hypertension (HTN).
2. Food Resources & Kitchen Skills (FoRKS), consisting of the same services as EUC plus home-delivered Mediterranean-style ingredient kits and virtual cooking classes for an additional 11 weeks with embedded lessons in kitchen organization, tool use, nutrition, budgeting, and shopping.

Assessments will be completed around Week 16 as the primary endpoint, and around Week 24 for maintenance evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English
2. Marion County resident
3. 35-75 years
4. Systolic BP of ≥120 in prior 12 months
5. Ability to see and read street signs (self report)
6. Stable housing with independent access to kitchen, including functional stove or hotplate, oven, refrigerator, and freezer (self report)
7. Activity independence per functional activities questionnaire (FAQ; <3 responses of "Require Assistance" and 0 responses of "Dependent")
8. Food insecurity per first two items of USDA 18-item survey with ≥ 1 response of "Often true" or "Sometimes true" [1) Within the past 12 months, you worried that your food would run out before you got the money to buy more; 2) Within the past 12 months, the food you bought just didn't last and you didn't have money to get more.] OR currently listed as food insecure in Eskenazi EMR; OR currently receiving SNAP benefits.
9. normal cognition per six-item screener (SIS; score of ≥ 5)
10. Mean systolic BP of ≥120 from 3 standard BP measurements taken by research staff following standardized wait periods.

Exclusion Criteria:

1. lives in nursing home
2. diagnosis of dementia or Alzheimer disease or mild cognitive impairment; Parkinson disease; brain tumor/infection/surgery (within the last 10 years with residual symptoms and/or functional loss/deficit, such as impaired learning, memory, or communication); psychosis, schizophrenia, or bipolar disorder
3. ICD 10 code I11/hypertensive heart disease, ICD 10 code I12/hypertensive CKD, ICD 10 code I13/hypertensive heart disease and CKD, ICD 10 code I15, or ICD 10 code I16
4. alcohol consumption ≥ 8 drinks per week for women, or ≥15 drinks per week for men
5. drug use/abuse (excluding marijuana) per EMR
6. moving out of area during study timeline
7. scheduling conflicts with intervention schedule
8. unwilling to use a touchscreen
9. unwilling to be on video conferencing
10. low communicative ability, functional status, or other disorders (examiner rated) that would interfere with interventions and assessments
11. unable to provide informed consent

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | End of treatment at Week 16
  Mean systolic blood pressure in FoRKS experimental arm compared to Enhanced Usual Care

SECONDARY OUTCOMES:
Hemoglobin A1c (HbA1c) | End of treatment at Week 16
  Mean hemoglobin A1c from blood in FoRKS experimental arm compared to Enhanced Usual Care

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O Clark, PhD, Principal Investigator — Indiana University; Richard Holden, PhD, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No